CLINICAL TRIAL: NCT04013360
Title: Acute Effect of Positive Expiratory Pressure Versus Breath Stacking Technique After Cardiac Surgery: a Randomized Crossover Trial
Brief Title: Acute Effect of Positive Expiratory Pressure Versus Breath Stacking Technique After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Prof. Dr. Antônio Marcos Vargas da Silva, Principal Investigator, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 92331518.6.0000.5346
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Complication, Postoperative; Cardiac Complication
Keywords: Cardiac Surgery; Positive End Expiratory Pressure; Physical Therapy Techniques; Pulmonary Funtcion
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breath Stacking (Active Comparator): Instrument composed of a one-way valve coupled to a face mask to promote the accumulation of successive inspiratory volumes.
  Interventions: Other: Breath Stacking; Other: Expiratory Positive Airway Pressure
- Expiratory Positive Airway Pressure (Active Comparator): Therapeutic technique consisting of a face mask, a one-way valve and an expiratory resistor, responsible for resistance to expiratory flow, which will determine the level of pressure in the airway.
  Interventions: Other: Breath Stacking; Other: Expiratory Positive Airway Pressure

INTERVENTIONS:
Other: Breath Stacking — The patients will perform the maneuver through successive inspiratory efforts for 20 s. Subsequently, the expiratory branch will be unobstructed to allow expiration. This maneuver will be repeated 5 times in each series, with intervals of 30 seconds between them. The technique will be performed with the trunk inclined 30º in relation to the horizontal plane, in 3 series, with interval of 2 min completing 15 min of therapy.
Other: Expiratory Positive Airway Pressure — Patients will perform exhalation of air through a facial mask containing an extrinsic positive expiratory pressure valve with a defined load of 10 cmH2O for 5 min. During the application of the technique the patients will have a trunk inclined 30º and will be stimulated to breathe normally, without effort or deep and fast breaths.

SUMMARY:
This study evaluates the efficacy and safety of a single session of positive expiratory pressure and of breath stacking technique in patients after cardiac surgery. The same patients will receive the two interventions, with an interval of 24 hours, and the acute effect of each will be verifed.

DETAILED DESCRIPTION:
Physiotherapy uses techniques and equipment that reduce postoperative pulmonary complications. The technique called breath stacking consists of an instrumental feature composed of a unidirectional valve coupled to a face mask to promote the accumulation of successive inspiratory volumes. The technique is used to prevent atelectasis and improve gas exchange. Another therapy is called expiratory positive airway pressure (EPAP) that uses positive end expiratory pressure (PEEP) in spontaneously breathing patients, keeping the airway open during expiration. The EPAP system consists of a face mask, a one-way valve and the expiratory resistor, which is responsible for resistance to expiratory flow, which will determine the level of PEEP.

ELIGIBILITY:
Inclusion Criteria:

Patients with indication for coronary artery bypass grafting and valve replacement, with surgical procedure for median sternotomy.

Exclusion Criteria:

* incapacity to understand the Informed Consent Form.
* cognitive dysfunction that prevents the performance of evaluations or interventions,
* intolerance to the use of EPAP or BS mask
* with chronic obstructive pulmonary disease (COPD)
* cerebrovascular disease
* chronic-degenerative musculoskeletal disease
* chronic infectious disease
* in treatment with steroids, hormones or cancer chemotherapy
* hemodynamic complications (arrhythmia, myocardial infarction during the operation, with blood loss ≥ 20% of the total blood volume, defined by Mannuci, et al., 2007)
* mean arterial pressure <70 mmHg and reduced cardiac output, requiring the use of intra aortic balloon or vasoactive drugs
* tracheal intubation for more than 12 hours after admission to the ICU or reintubated
* individuals unable to maintain airway permeability.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Tidal volume | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  It will be evaluated preoperatively and also before and after 10 minutes of each intervention, in the postoperative period. This measurement will be obtained through the the division of the minute volume by the respiratory rate.
Forced vital capacity (FVC) | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  It will be evaluated preoperatively and also before and after 10 minutes of each intervention, in the postoperative period, as recommended by the American Thoracic Society and European Respiratory Society (2006) and based on reproducibility and acceptability criteria, three maneuvers will be performed (variability <5%) and considered the best curve for the study.

SECONDARY OUTCOMES:
Forced expiratory volume in the first second (FEV1) | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  It will be evaluated preoperatively and also before and after 10 minutes of each intervention, in the postoperative period, as recommended by the American Thoracic Society and European Respiratory Society (2006) and based on reproducibility and acceptability criteria, three maneuvers will be performed (variability <5%) and considered the best curve for the study.
Peak expiratory flow (PEF) | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  It will be evaluated preoperatively and also before and after 10 minutes of each intervention, in the postoperative period, as recommended by the American Thoracic Society and European Respiratory Society (2006) and based on reproducibility and acceptability criteria, three maneuvers will be performed (variability <5%) and considered the best curve for the study.
Forced expiratory flow between 25 and 75% of the curve of FVC (FEF25-75) | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  It will be evaluated preoperatively and also before and after 10 minutes of each intervention, in the postoperative period, as recommended by the American Thoracic Society and European Respiratory Society (2006) and based on reproducibility and acceptability criteria, three maneuvers will be performed (variability <5%) and considered the best curve for the study.
Minute volume | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  It will be evaluated preoperatively and also before and after 10 minutes of each intervention. To obtain the Minute Volume (MV), the patient will be instructed to inhale and exhale slowly for one minute and the value of MV and respiratory rate (RR) will be recorded. The respiratory rate was measured by the movements of the rib cage during respiratory cycles performed in one minute. The MV will be obtained by a Wright ® ventilometer (British Oxigen Company, London, England).
Respiratory rate | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  They will be assessed at baseline, immediately after and 10 minutes after each intervention. The respiratory rate was measured by the movements of the rib cage during respiratory cycles performed in one minute.
Heart rate | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  They will be assessed at baseline, immediately after and 10 minutes after each intervention, through multi-parameter monitor.
Peripheral Oxygen Saturation (SpO2) | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  They will be assessed at baseline, immediately after and 10 minutes after each intervention through the G-Tech® portable pulse oximeter.
Blood pressure | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  They will be assessed at baseline, immediately after and 10 minutes after each intervention. The blood pressure will be obtained through multi-parameter monitor.
Heart work measurement | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  They will be assessed at baseline, immediately after and 10 minutes after each intervention through the calculation of the double product (multiplication of systolic blood pressure by heart rate).
Thoracoabdominal mobility | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  Will be evaluated by thoracic and abdominal cirtometry
Painful perception in the surgical incision | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  Will be assessed at baseline, immediately after and 10 minutes after each intervention through a Visual Analog Scale, a one-dimensional instrument for evaluation of pain intensity, with a range of 1 to 10.
Degree of dyspnea | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  Will be assessed at baseline, immediately after and 10 minutes after each intervention, through the Modified Borg Scale, a vertical scale quantified from 0 to 10. Zero represents no symptoms and 10 represents maximum symptoms.
Signs of respiratory discomfort (dizziness, tachypnea, sweating, use accessory musculature) | 12 to 24 hours after removal of drains and 24 hours after primary intervention
  They will be assessed at baseline, immediately after and 10 minutes after each intervention, through clinical inspection.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Santa Maria, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided